CLINICAL TRIAL: NCT02991547
Title: Study on Outcomes of Active Surveillance Among Invasive Locoregional Adenocarcinoma of Esophagus and Gastroesophageal Junction (GEJ) With Complete Response After Neoadjuvant Combined Chemoradiotherapy
Brief Title: Surveillance of Patients With Adenocarcinoma of the Gastroesophageal Junction or Esophagus
Acronym: SAGE
Status: Terminated | Type: Observational
Why Stopped: Initial Principal Investigator no longer at institution.
Sponsor: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 1611-55
Record Dates: First submitted 2016-11-28; First posted 2016-12-13 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Adenocarcinoma Esophagus
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observational

SUMMARY:
The purpose of this study is to find out more information about patients who have cancer (adenocarcinoma) of the esophagus or gastroesophageal junction (GEJ) who have been treated with chemotherapy and radiation but have not had surgery. The study will follow patients for 5 years to monitor for their cancer and to see how the standard medical care affects the daily life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of esophagus or gastroesophageal junction (nidus of the cancer within 5 cm from the gastroesophageal junction) confirmed by biopsy with clinical stage I, II, or III. The superficial adenocarcinoma of the esophagus will be excluded.
* Received no previous treatment for esophageal cancer.
* Measurable or evaluable disease
* ECOG performance status: 0 to 2 that is able to perform activities of daily living with minimal assistance
* Adequate bone marrow function (hemoglobulin ≥8 g/dl, neutrophil ≥1.5x109/L and platelet ( ≥100x109/L)
* Adequate liver function

  * Bilirubin normal, Meets 1 of the following criteria:
  * Alkaline phosphatase (AP) normal AND AST/ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST/ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST/ALT normal
* Adequate kidney function (creatinine ≤1.5 UNL and creatinine clearance ≥ 60 )
* Be at least 4 weeks from recent major surgical procedures.
* Patients must be able to understand the nature of the study and give written informed consent
* At least one measurable lesion on CT, MRI or esophageal barium exam.

Exclusion Criteria:

* Age < 18 years and >80 years
* Contraindication for irradiation: complete obstruction of esophagus, deep esophageal ulcer, fistula to mediastinum, or hematemesis
* Participating in other clinical trials
* Pregnancy
* Clinically significant and uncontrolled major medical conditions including but not limited to active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia, psychiatric illness/ social situation that would limit compliance with study requirements
* any medical condition, which in the opinion of the study investigator places the subject at an unacceptably high risk for toxicities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adenocarcinoma of the esophageal and gastroesophageal junction
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2016-12; Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
Rate of complete remission | 8 weeks after completion of neoadjuvant chemoradiotherapy
Occurrence of local recurrence or mestastasis or both | 5 years
Adverse effect profile | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joyson Poulose, MD, Study Director — Guthrie Medical Group, PC/Robert Packer Hospital
Locations (2):
- United States (2):
  - Guthrie Corning Hospital, Corning, New York
  - Guthrie Medical Group, PC/Robert Packer Hospital, Sayre, Pennsylvania

IPD SHARING:
Plan to Share IPD: No